CLINICAL TRIAL: NCT01375855
Title: Late Incomplete Stent Apposition Evaluation II: Vascular Effects Evaluation After Polimer and No-polimer Based Coronary Artery Drug Eluting Stent Ilmplantation. An IVUS Based Study
Brief Title: Late Incomplete Stent Apposition Evaluation II: Comparison Between Polimer-based and No-polimer Stent System. IVUS Based Study
Acronym: LISAII
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Unitat de Hemodinàmic. Servei Cardiologia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-000142-12
Record Dates: First submitted 2010-12-28; First posted 2011-06-17 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2007-02

CONDITIONS: Coronary Artery Disease
Keywords: Late stent malapposition; stent thrombosis; IVUS; non-polimeric stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Angioplasty, Balloon, Coronary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polimeric-PES (Active Comparator): Arm receiving polimeric stent (Taxus)
  Interventions: Procedure: Percutaneous transluminal Coronary Angioplasty
- Non-Polimeric PES (Active Comparator): Arm receiving non-polimeric PES (axxion)
  Interventions: Procedure: Percutaneous transluminal Coronary Angioplasty

INTERVENTIONS:
Procedure: Percutaneous transluminal Coronary Angioplasty — Coronary artery stent implantation

SUMMARY:
Vascular effects evaluation after non-polimeric and polimeric paclitaxel stent implantation.In particular the investigators will use Taxus )as a polimeric stent)and Axxion (as a non-polimeirc)stent system. The investigators will look at late stent malapposition by means of intracoronary ultrasound imaging technique (IVUS) at baseline and 9 months follow-up. The investigators sought to compare the two stent types with the same drug to verify the polimer role. The polimer itself seems to provoke inflammation and hypersensibility if the arterial wall and it seems to be the base of a process of positive remodeling found at drug eluting stent implantation site.

This positive remodeling is the mechanism producing late stent malapposition which on its turn can determine stent thrombosis, as demonstrated by pathological studies. At the same time the investigators will study the incidence of clinical events like myocardial infarction, stent thrombosis, TLR and death along with the incidence of angiographic restenosis at 2 years follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery stenosis in one, two or three vessels, and with objective evidence of isquemia.
* The stenosis must allow IVUS analisis, must be treatable with angioplasty with stent
* Target Vessel diameter must be between 2.25- 4 mm with QCA.
* Patients must sign informed consent
* Patients and their physician must accept the angiographic follow-up

Exclusion Criteria:

* 18 years old patients
* SCA within the last 72 hours, or patients with CK twice over the upper normal limit
* Pregnancy
* Target vessel diameter < 2.25 or > 4 mm by QCA
* Previous brakitherapy or DES in the target lesion
* Restenotic lesion
* -Allergy to aspirin, clopidogrel or ticlopidin
* Patients enrolled in other studies or trials
* By-pass graft lesions
* Real bifurcationa lesions
* Severe Renal insufficiency (creatinin clearance < 30 ml/min).
* Severe Liver failure(GOT y GPT > 3 times the upper normal limit)
* Life expectancy < 1 year because of other pathologies

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2007-10

PRIMARY OUTCOMES:
Intra coronary ultrasound analysis to verify stent malapposition at follow-up | 9 months

SECONDARY OUTCOMES:
Clinical events (myocardial infarction, TLR,at 1, 9, 12, 24 months follow-up:; Incidence of restenosis with QCA at 9 months follow-up Intimal hiperplasia measured by IVUS at 9 months follow-up; Stent Thrombosis. | 9 months and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Manel Sabate, MD, PhD, Principal Investigator — Hospital de la Santa Creu Y Sant Pau, Unidad de Hemodinamica
Locations (1):
- Hospital de la Santa Creu y Sant Pau, Barcelona, Spain, Spain

REFERENCES:
- [Background] Hong MK, Mintz GS, Lee CW, Park DW, Lee SW, Kim YH, Kang DH, Cheong SS, Song JK, Kim JJ, Park SW, Park SJ. Impact of late drug-eluting stent malapposition on 3-year clinical events. J Am Coll Cardiol. 2007 Oct 9;50(15):1515-6. doi: 10.1016/j.jacc.2007.07.038. Epub 2007 Aug 27. No abstract available. PMID 17919574
- [Derived] Shiratori Y, Cola C, Brugaletta S, Alvarez-Contreras L, Martin-Yuste V, del Blanco BG, Ruiz-Salmeron R, Diaz J, Pinar E, Marti V, Garcia-Picart J, Sabate M. Randomized comparison between polymer-free versus polymer-based paclitaxel-eluting stent: two-year final clinical results. Circ Cardiovasc Interv. 2014 Jun;7(3):312-21. doi: 10.1161/CIRCINTERVENTIONS.113.000800. Epub 2014 May 6. PMID 24803435